CLINICAL TRIAL: NCT02930460
Title: Prospective Cohort Study of Patients Intolerant to High Pressure Under Continuous Positive Airway Pressure, Treated With Bilevel Positive Airway Pressure (AirCurve 10 VAutoTM) as Second-line Therapy: PoP IN VAuto
Brief Title: Prospective Cohort Study of Patients Intolerant to High Pressure Under Continuous Positive Airway Pressure Treated With Bilevel Positive Airway Pressure as Second-line Therapy.
Acronym: PoP IN VAuto
Status: Terminated | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: PoP IN VAuto
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2017-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective observational study of obstructive Sleep Apnea patients treated with Bilevel Positive Airway Pressure: AirCurve 10 VAutoTM

DETAILED DESCRIPTION:
To characterize, in routine practice, non compliant patient to continuous positive airway pressure who can get a benefit of a bilevel positive airway pressure therapy as a second line treatment (Aircurve 10 VAutoTM ) To evaluate the clinical management of obstructive sleep apnea patients treated by Aircurve 10 VAutoTM , especially impact on compliance and residual apnea hypopnea Index.

To evaluate Aircurve 10 VAutoTM benefit on quality of Life and quality of sleep

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Obstructive Sleep Apnea Patient previously treated by Continuous positive airway pressure non-compliant to therapy
* Patient naive of bilevel Positive Airway Pressure therapy

Exclusion Criteria:

* Bilevel positive airway pressure Contraindication
* Severe respiratory disease diagnostic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obstructive sleep apnea patient, non compliant or intolerant to Continous positive Airway Pressure therapy, treated by Bilevel Positive Airway Pressure (Aircurve 10 VAutoTM ) as second line therapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-11; Primary Completion 2018-11 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Compliance | 3 months
  hours of usage of the device per night

SECONDARY OUTCOMES:
sleepiness | 3 months
  Epworth sleepiness score evolution
sleep quality | 3 months
  Pittsburgh sleep questionnaire index

CONTACTS AND LOCATIONS:
Overall Officials: Alain Palot, MD, Principal Investigator — CHU Marseille
Locations (8):
- France (8):
  - CH de Belfort, Belfort
  - Clinique Aguilera, Biarritz
  - Cabinet de Pneumologie, Blois
  - HCL - Croix-Rousse Hospital, Lyon
  - APHM, Marseille
  - Centre médical du sommeil, Metz
  - Hopital Saint Antoine, Paris
  - Polyclinique Saint-Laurent, Rennes

IPD SHARING:
Plan to Share IPD: No